CLINICAL TRIAL: NCT04759781
Title: A Prospective Registry Study of a Primary Melanoma Gene-signature to Predict Sentinel Node (SN) Status and Determine Its Prognostic Value for More Accurate Staging of SN-negative Melanoma Patients.
Brief Title: MElanoma Research Lymph Node Prediction Implementation National_001
Acronym: MERLIN_001
Status: Active, not recruiting | Type: Observational
Sponsor: SkylineDx (Industry)
Responsible Party: Sponsor
Other Study IDs: MERLIN_001
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Melanoma
Keywords: prospective study; gene expression; melanoma; Merlin; assay
MeSH Terms: conditions — Melanoma; Neurofibromatosis 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
MERLIN_001 is a prospective registry study of a primary melanoma gene-signature to predict sentinel node (SN) status and to determine its prognostic value for more accurate staging of SN-negative melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with invasive malignant melanoma of the skin (AJCC 8th edition staging guidelines) elected to undergo sentinel lymph node biopsy per the treating physician's recommendation.
* Male or female, age ≥18 years.

Exclusion Criteria:

* Full primary melanoma pathology report unavailable.
* Documented clinically apparent nodal metastases at diagnosis.
* Distant metastatic disease (M1a,b,c,d) clinically present at primary diagnosis
* Any prior or concurrent primary invasive melanoma mapping to the same draining lymph node basin(s).
* Documented history of another (prior or concurrent) primary invasive melanoma of T1b or greater at any site within the last 5 years.
* Previous surgery in or radiation therapy to the draining lymph node basin(s) of the current primary melanoma.
* Ocular, vulvar, perianal or mucosal melanomas or melanocytic tumors of uncertain malignant potential (MELTUMP) or atypical Spitz tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospectively collected primary cutaneous melanoma patients who are elected per treating physician's recommendation to undergo sentinel lymph node biopsy.
Sampling Method: Probability Sample
Enrollment: 1820 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Negative Predictive Value (NPV) | 2 years after inclusion
  The predictive capability of the Merlin Assay to identify newly diagnosed primary cutaneous melanoma patients who have a low risk of presenting with a positive sentinel lymph node.
Positive Predictive Value (PPV) | 2 years after inclusion
  The predictive capability of the Merlin Assay to identify newly diagnosed primary cutaneous melanoma patients who have a low risk of presenting with a positive sentinel lymph node.
Sensitivity and Specificity. | 2 years after inclusion
  The predictive capability of the Merlin Assay to identify newly diagnosed primary cutaneous melanoma patients who have a low risk of presenting with a positive sentinel lymph node.

SECONDARY OUTCOMES:
3-5 year Recurrence-Free Survival (RFS) | 3-5 years after patient inclusion
  Time between the date of sentinel lymph node biopsy procedure and the date of first melanoma recurrence (loco-regional or distant metastasis) or date of death (whatever the cause), whichever occurs first.
3-5 year Distant Metastasis-Free Survival (DMFS) | 3-5 years after patient inclusion
  Time between the date of sentinel lymph node biopsy procedure and the date of first distant metastasis or date of death (whatever the cause), whichever occurs first.
3-5 year Overall Survival (OS) | 3-5 years after patient inclusion
  Time between the date of sentinel lymph node biopsy procedure and the date of death (whatever the cause).

CONTACTS AND LOCATIONS:
Overall Officials: Vernon K. Sondak, MD, Principal Investigator — Moffitt Cancer Center; Tina J. Hieken, MD, Principal Investigator — Mayo Clinic; Michael E. Egger, MD, MPH, Principal Investigator — University of Louisville
Locations (9):
- United States (9):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No